CLINICAL TRIAL: NCT03800459
Title: Effect of a Family Empowerment Program on Coping With Stress, Problem Solving in Parents, and Quality of Life in Children With Cystic Fibrosis: Randomized Controlled Trial
Brief Title: Effect of a Family Empowerment Program on Coping, Problem Solving in Parents, and Quality of Life in Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Fatma Taş Arslan, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-4242
Record Dates: First submitted 2018-12-28; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
Keywords: Children with Cystic Fibrosis; Parents; Quality of Life; Coping with Stress; Problem Solving; family empowerment program; Nursing
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blindness in the study was done by data collectors and statisticians. The data were collected by the nurse who did not know who is in the experiment and control group.
  To reduce selection bias and to control the variables that may have an effect on outcome variables, random assignment was made to the experimental and the control group by a statistician who did not know the names and characteristics of the parents of and children with CF. The analysis of the data coded according to the groups was made by a statistician. After the statistical analyses were completed and the research report was written, the researcher explained the coding for the experimental and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention group (Experimental): Experimental: Intervention group
  Interventions: Behavioral: family empowerment program
- Control:no intervation group (No Intervention): Control:no intervation group

INTERVENTIONS:
Behavioral: family empowerment program — The empowerment program-nursing interventions were given in 6 sessions in the experimental group Session 1: Individualized training: General information about CF, respiratory system involvement and treatment process, airway cleaning in CF, drug applications (45-50 min) Session 2:Phone calls: Motivational and reminder interviews were carried out in order to reinforce the content of the first individual training (15 min).Session 3:Phone calls:Motivational and reminder interviews were carried out in order to reinforce the content of the first individual training (15 min) Session 4:Individualized training:protection from infections, nutrition and psychosocial support (45 min) Session 5:Phone calls: Motivational and reminder interviews were carried out in order to reinforce the content of the second individual training. (10 min) Session 6:Phone calls: Motivational and reminder interviews were carried out in order to reinforce the content of the second individual training. (10 min)
  Arms: Experimental: Intervention group

SUMMARY:
Parents of children with cystic fibrosis (CF) experience high levels of stress and problems. Family empowerment interventions provide important support for many patients with CF and their families. However,there is a lack of research exploring the effects of such empowerment programs on coping, and Problem Solving among parents, and Quality of Life in Children with CF.

The present study aimed to assess the effect of a family empowerment program-based nursing intervention on parents coping with stress and problem solving, and quality of life children with CF.

DETAILED DESCRIPTION:
Parents of children with cystic fibrosis (CF) experience high levels of stress and problems. Family empowerment interventions provide important support for many patients with CF and their families. However,there is a lack of research exploring the effects of such empowerment programs on coping, and Problem Solving among parents, and Quality of Life in Children with CF. The present study aimed to assess the effect of a family empowerment program-based nursing intervention on parents coping with stress and problem solving, and quality of life children with CF.

A single-blinded, parallel group pretest and posttest design randomized controlled trial was used.

Data were collected over 5 months (January 2017-May 2017) from 48 participants in a medical faculty hospital. They were randomly assigned to the experimental (n = 24) and control (n = 24) groups. Nursing interventions applied to the experimental group for ten weeks with the intent of strengthening families consist of; providing individualized training and booklet concerning disease management and providing phone calls and consultancy services for the purpose of reinforcing the training and increasing the motivation. A routine polyclinic follow-up was applied to the control group. Problem Solving Inventory (PSI), Scale of Ways of Coping with Stress (SWCS), and The Cystic Fibrosis Questionnaire-Revised scale (CFQ-R) were used reliable and valid instruments. The data were evaluated using the Wilcoxon Signed Ranks test in evaluating dependent groups and the Mann-Whitney U test in independent groups.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-18 years old;
* Pulmonary functions Forced Expiratory Volume (FEV 1) over 40%
* being able to communicate in Turkish,
* voluntary parents in the study.

Exclusion Criteria:

* had mental disorders;
* receiving mechanical ventilation;
* Being in the process of lung transplantation;
* having a sister/brother who died due to CF
* Being in enteral or parenteral feeding;
* having a chronic disease other than CF.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2017-02-26 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Child and parents information form | 3 weeks
  The form was developed to define baseline characteristics and was based on previous literature. The questionnaire included questions regarding the sociodemographic characteristics of the participants, such as age, gender, educational level, income, duration of treatment and diagnosis.

SECONDARY OUTCOMES:
Problem Solving Inventory (PSI) | 10 weeks
  Problem Solving Inventory (PSI) was measured using the 35-item Problem Solving Inventory Scale (Heppner & Petersen, 1982). PSI; is a 35-item measure with a six-point Likert scale that assesses an individual's perceptions of his or her problem-solving styles, rather than actual problem-solving skills. Higher scores indicate an individual's assessment of oneself as a relatively ineffective problem solver. The PSI has a total score derived from three scales. The three subscales are: (a) Problem-Solving Confidence (PSC, 11 items); (b) ApproachAvoidance Style (AAS, 16 items); and (c) Personal Control (PC, 5 items). The PSC refers to an individual's belief and trust in one's own problem-solving ability. The AAS is defined as a general tendency to approach or avoid a wide range of problem-solving activities. The PC refers to individual's belief that one is in control of his or her own behaviors and emotions while solving problems.
Scale of Ways of Coping with Stress (SWCS) | 10 weeks
  The SWCS was developed by Folkman and Lazarus in 1980 (Folkman & Lazarus 1980). The Turkish adaptation and validity study of SWCS was conducted by Şahin and Durak in 1995 (Şahin & Durak 1995). The SWCS is a 4-point Likert-type scale ranging from 1 (Not appropriate) to 4 (Very appropriate). In the Turkish adaptation and validity study of the SWCS, factor analysis, comparisons of measurement-correlating validity and counter groups and validity for the SWCS were conducted and Cronbach's alpha reliability coefficients of the subscales were found between 0.45 and 0.80. The scale consisted of two groups; one was the effective coping ways (ECWs), which contained the optimistic approach, self-confident approach, and seeking social support, and the other group was the ineffective coping ways (ICWs), which included the hopelessness and submissive approaches.
The Cystic Fibrosis Questionnaire-Revised (CFQ-R) | 10 weeks
  The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a CF-specific health-related quality of life (HRQOL) questionnaire (Quiitner et al. in 2005). The CFQ-R is a 4-point Likert-type scale ranging from 1 to 4. Higher scores indicate better HRQOL

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Tas Arslan, Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Donmez H, Tas Arslan F. The Effectiveness of a Parent Empowerment Intervention for Caregivers of Children with Cystic Fibrosis: A Randomized Controlled Trial. Compr Child Adolesc Nurs. 2024 Dec;47(4):267-283. doi: 10.1080/24694193.2024.2411986. Epub 2024 Oct 9. PMID 39382937